CLINICAL TRIAL: NCT07059247
Title: Periodontal Regeneration at the Distal Site of Second Molars After the Extraction of Lower Included Third Molars
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23/308-EC_X
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Tooth Extraction; Wisdom Tooth Removal; Periodontal Regeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Application of EMD after the extraction
  Interventions: Biological: Application of Enamel Matrix Derivatives; Procedure: Extraction of the impacted third molar
- Control (Sham Comparator): No application of EMD after the extraction
  Interventions: Procedure: Extraction of the impacted third molar

INTERVENTIONS:
Biological: Application of Enamel Matrix Derivatives — After the extraction of the impacted lower third molar, EMD will be applied on the distal site of the second molar
  Arms: Test group
Procedure: Extraction of the impacted third molar — Extraction of the impacted third molar

SUMMARY:
From an exclusively periodontal point of view, the extraction of third molars (3M) or wisdom teeth is relatively frequently recommended, either because they show reduced bone support or to avoid periodontal damage to the supporting bone of the adjacent second molar (2M). There are anatomical conditions that make plaque control difficult for the patient, and it is common to find periodontal pockets with significantly increased depths on the distal side of second molars that are or have been closely associated with an impacted third molar.

Among the periodontal considerations regarding impacted third molars, two aspects have traditionally been included: 1)The periodontal damage that certain impactions can cause to the periodontal health of the second molar, and 2) the periodontal sequelae or complications that the extraction of a wisdom tooth may leave on the distal surface of that second molar.

Various therapeutic approaches have been described in the literature to prevent periodontal damage following the surgical intervention involved in the extraction of a fully or partially impacted wisdom tooth. These include scaling of the distal surface of the 2M after extraction, modifications in the surgical technique - such as flap design or suturing method - and various regenerative techniques.

Within this context, the clinical research in which we invite the patients to participate will be developed. We will study the changes in bone levels on the posterior part of the second molar that is in contact with or close to the third molar, as well as the health of the soft tissues, after performing a conventional extraction protocol of the impacted lower third molar. This protocol includes the placement of a regenerative material of porcine origin (test procedure; enamel matrix derivatives) and will be compared to extraction without such material - and therefore without any attempt at periodontal regeneration (standard procedure). The patients will be closely followed up to one year after the surgical performance. This follow-up will be performed clinically and radiographically.

ELIGIBILITY:
Inclusion Criteria:

* Adult (< 18 years old) patients with impacted or semi-impacted lower third molars and with indication of extraction
* Systemically healthy patients
* Non-smokers or less than 10 cigarettes per day

Exclusion Criteria:

* Patients with uncontrolled systemic diseases (ASA III-IV)
* Medication that potentially affects bone metabolism
* Absence of adjacent lower second molar
* Presence of crowns, distal caries or distal fillings of the adjacent second molar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level | From enrollment to the end of treatment at 1 year

SECONDARY OUTCOMES:
Pocket Probing Depth | From enrollment to the end of treatment at 1 year
Radiographic Bone Level Changes | From enrollment to the end of treatment at 1 year